CLINICAL TRIAL: NCT01869400
Title: An Observational, Multicenter, Open-label Study of YONDELIS®+PLD for the Treatment of Patients With Platinum-sensitive Relapse of Ovarian Cancer
Brief Title: An Observational Study of YONDELIS®+PLD for the Treatment of Patients With Platinum-sensitive Relapse of Ovarian Cancer
Acronym: NIS-OvaYond
Status: Completed | Type: Observational
Sponsor: PharmaMar, Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: OvaYond
Record Dates: First submitted 2013-05-15; First posted 2013-06-05 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Yondelis-Pegylated liposomal Doxorubicin: 30 mg/m² PLD i.v. followed by 1.1 mg/m² Yondelis® i.v. 3 h, q3weeks

SUMMARY:
Clinical trials are, due to the inclusion and exclusion criteria, accomplished with defined patient groups, which are not representative for the whole patient population.

Especially elderly patients and patients with co-morbidities are underrepresented in clinical trials.

This non-interventional study will examine the efficiency and toxicity of the Yondelis® + PLD combination therapy in a general patient population to evaluate if the data collected in the clinical trials can be assigned to a general patient population.

DETAILED DESCRIPTION:
Yondelis® (trabectedin) was approved (in combination with PLD) in the European community in December 2009 for the treatment of platinum-sensitive ovarian cancer relapse. Based on the outcomes of study OVA-301, this non-interventional study will investigate the role of a platinum-free treatment regimen in patients with progressive ovarian cancer relapsing > 6 months after completing previous platinum-based chemotherapy. In particular, this study aims at collecting the "real-life" data with regard to the response and the influence of the mentioned therapy on the "tumor related events", to objectify the value of palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Women age >18, no upper limit
* Patients with relapsed platinum-sensitive ovarian cancer
* Before inclusion in the NIS written informed consent must be given

Exclusion Criteria:

* According to summary of product characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitales and medical practices in Germany
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
safety and tolerability data of the study therapy | during Yondelis-PLD-therapy
  Number of patients with adverse events

SECONDARY OUTCOMES:
"Real life data" - clinical and / or serological (CA 125) response and Stable disease rates | till one year after last date of Yondelis-PLD-therapy
  Number of patients with CR, PR, SD as best response
Treatment duration | during Yondelis-PLD-therapy
  Time between first and last cycle of each patient
Observation of the number of the therapy cycles applied | during Yondelis-PLD-therapy
  Number of applied therapy cycles
Time to next treatment | 1 Year after last Yondelis-PLD-Therapy
  Date from last Yondelis-PLD-treatment to date of next treatment
Progression free survival | till one year after last date of Yondelis-PLD-therapy
  Difference between date of first documentation of "PD" and the date of first Yondelis® + PLD application
Duration of response | till one year after last date of Yondelis-PLD-therapy
  Time in months from first assessment of CR or PR until the first date of PD or death.

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Runnebaum, Prof. Dr., Study Chair — Klinikum der Friedrich-Schiller-Universität Jena, Klinik für Frauenheilkunde, Bachstr. 18, D-07743 Jena
Locations (2):
- Germany (2):
  - Praxis und Tagesklinik für gynäkologische Onkologie, Ebersberg, Bavaria
  - Diakoniekrankenhaus, Gynäkologie und Geburtshilfe, Rotenburg (Wümme), Lower Saxony

IPD SHARING:
Plan to Share IPD: Undecided